CLINICAL TRIAL: NCT03142906
Title: Perioperative Point-of-Care Ultrasound: A Randomized Controlled Trial
Brief Title: Perioperative Point-of-Care Ultrasound
Acronym: POCUS-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Ahmed Hegazy, Assistant Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 108613
Record Dates: First submitted 2017-04-28; First posted 2017-05-08 (Actual); Last update posted 2018-07-16 (Actual); Status verified 2018-07

CONDITIONS: Anesthesia; Ultrasound; Emergencies; Operation; Ultrasonography; Surgery
Keywords: preoperative, perioperative, point-of-care ultrasound
MeSH Terms: conditions — Emergencies | interventions — Radionuclide Imaging

STUDY DESIGN:
Intervention Model Description: Randomized parallel group controlled clinical trial
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor blinded to patient assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scan group (Experimental): Patients randomized to the scan group (intervention arm) will receive a preoperative point-of-care ultrasound (POCUS) exam as an adjunct to their preoperative assessment, the results of which will be disclosed to the anesthesiologist and the patient care team. This POCUS exam will include a focused cardiac ultrasound, a lung and pleural ultrasound, and a gastric volume and content ultrasound assessment. Patients randomized to this arm may also receive repeat POCUS exams as needed and as clinical conditions change. These repeat exams may be requested by the anesthesiologist or patient care team.
  Interventions: Diagnostic Test: Scan
- No scan group (No Intervention): Patients randomized to no scan (control arm) will not receive a preoperative point-of-care ultrasound exam. Patients in this arm will receive the standard-of-care; a routine preoperative assessment and physical examination by their attending anesthesiologist.

INTERVENTIONS:
Diagnostic Test: Scan — The preoperative point of care ultrasound includes a protocolized focused cardiac ultrasound, lung and pleural ultrasound and a gastric volume and content ultrasound assessment, all of which will be performed as an adjunct to the anesthesiologist's assessment. The result of this ultrasound examination will be disclosed to the anesthesiologist and patient care teams. Repeat ultrasounds may be done as the patient's clinical condition changes, or as requested by the anesthesiologist or patient care team.
  Other Names: POCUS; Ultrasound examination; Point-of-care ultrasound
  Arms: Scan group

SUMMARY:
The goal of this study is to assess the impact of perioperative point-of-care ultrasound (POCUS) assessment on patient-important outcomes (e.g. hospital length of stay, length of stay in recovery, mortality etc.) and perioperative patient management strategies, in patients undergoing non-elective non-cardiac surgeries.

DETAILED DESCRIPTION:
Preoperative patients undergoing emergency non-cardiac surgery will be approached for study recruitment and participation. Study participants will be randomized to receive, or not, a preoperative POCUS exam as part of their routine preoperative assessment. Patients randomized to receiving a POCUS exam will undergo a protocolized focused cardiac ultrasound, lung and pleural ultrasound and a gastric volume and content ultrasound assessment. Results of this exam will be disclosed to the anesthesiologist and primary care team. Randomization will be stratified by the presence of any sign(s) of cardiorespiratory failure. Signs of cardiorespiratory failure are defined as: systolic blood pressure <90 mmHg, heart rate>100, respiratory rate >24, Oxygen saturation <90%, requirement of supplemental oxygen or mechanical ventilation, new requirement of loop diuretics in current hospital admission, chest pain, newly diagnosed ECG changes, requirement of vasoactive drugs, signs of pre-renal azotemia (BUN:creatinine ratio >20). Outcome data will be collected prospectively. Investigators performing and interpreting the scan will disclose the results to the care team but will not participate in patient care. Primary and secondary outcome data collection will be performed by an investigator blinded to patient assignment. The primary outcome is post anesthetic care unit length-of-stay. The secondary outcomes are post-randomization hospital length of stay, number of operating room (OR) delays for optimization, alterations in anesthetic management (using a brief anesthesiologist-administered survey), intensiveness of OR management (invasive blood pressure monitoring, central venous pressure monitoring, intraoperative TEE), new peri-operative diuretic use, new intensive care admission rates, mortality during this admission, amount/frequency of postoperative investigations, rates of detection of new pathologies identified by preoperative POCUS exam and the rates of adequately diagnostic POCUS studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >17 years
* Undergoing urgent or emergent non-cardiac surgery classified as intermediate or high risk according to American Heart Association(AHA)/American College of Cardiology(ACC) guidelines.

These include vascular surgeries (supra or infra-inguinal), intraperitoneal surgeries, intra-thoracic surgeries, head and neck surgeries, spine surgeries, urologic surgeries, and proximal extremity orthopedic surgeries. Peripheral extremity surgeries (wrist or below, and ankle or below), in addition to appendectomies and cholecystectomy surgeries will be excluded from this study.

Exclusion Criteria:

* Patients scheduled for elective or pre-booked surgeries
* Patients undergoing cardiac surgeries
* Patients undergoing low risk procedures e.g. endoscopic procedures, superficial skin, subcutaneous tissue, breast, ophthalmic, and ambulatory surgeries
* Patients undergoing orthopedic peripheral extremity surgeries (e.g. ankle, wrist, hand, foot)
* Patients who have had an echo during the current hospital admission prior to recruitment.
* Patients where the investigator performing or over-reading the POCUS scan is required to participate directly in perioperative patient care (e.g. anesthesiologist co-investigator performing or over-reading scan is on-call for this emergency case)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2017-04-04 (Actual); Primary Completion 2018-08-01 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Post-anaesthesia care unit (PACU) length of stay | From time of PACU admission until the time of transfer from PACU, assessed up to 48 hours.
  Total time (minutes) from postoperative PACU admission to PACU discharge.

SECONDARY OUTCOMES:
Post-randomization hospital length-of-stay | From date of randomization until the date of hospital discharge or death from any cause, whichever came first, assessed up to 4 weeks.
  Number of days in hospital from study enrollment to discharge or death.
New ICU admission rates | From time of randomization to the immediate postoperative period, assessed up to 6 hours after the conclusion of surgery.
  New admissions to ICU in the immediate post operative period in patients previously on the ward or in the emergency department.
Rates of detection of unexpected or new pathologies | From time of randomization to the time of interpretation of the last POCUS scan, assessed up to 2 weeks from randomization.
  New cardiac, pulmonary or gastric pathology detected by preoperative POCUS not known to be present previously. Examples include valve lesions, resting regional wall motion abnormalities, ventricular dysfunction, ventricular hypertrophy, pulmonary edema, consolidation and/or pleural effusion. This will be calculated only for participants randomized to the Scan Group.
Change in anesthetic plan based on the scan result | From time of randomization to the time of interpretation of the last POCUS scan, assessed up to 2 weeks from randomization.
  A survey will be administered to the anesthesiologist caring for the patient asking whether the POCUS exam findings influenced the anesthetic plan for the patient. If the answer is "yes, it did influence the anesthetic plan", subsequent questions will explore how it influenced anesthetic management. These will include questions of whether it influenced fluid management, anesthetic technique, choice of invasive lines, choice or dose of induction agents, or delay of surgery for optimization or further work-up. This will be calculated only in participants randomized to the Scan Group.
Intensiveness of operating room (OR) management | During OR time post randomization, assessed until the patient is transferred from the OR to PACU, up to 7 days from randomization.
  Use of invasive lines i.e. arterial, central lines or TEE monitoring
New or change in peri-operative diuretics use | From time of enrollment, up to 2 weeks from randomization.
  New use or change in pattern of diuretic use in the pre, intra or post operative phases.
Rates of blood work ordered and imaging investigations | From time of enrollment, up to 2 weeks from randomization.
  Frequency of post-randomization blood draws, frequency of post-randomization imaging studies (X-rays, CT's, MRI's, ultrasounds, echoes, and nuclear scans).
Mortality | From time of enrollment, up to 4 weeks from randomization.
  In-hospital post randomization mortality rate. Patients dying after transfer to another acute care hospital will also be counted as an in-hospital post randomization mortality.
Rates of adequately diagnostic focused cardiac ultrasounds, lung and pleural ultrasounds, and gastric volume/content assessments. | From time of randomization to the time of interpretation of the last POCUS scan, assessed up to 2 weeks from randomization.
  An adequately diagnostic focused cardiac ultrasound will be defined as a scan having two or more views showing at least 3 cardiac chambers with diagnostic quality. An adequately diagnostic lung and pleural scan will demonstrate a clear aeration pattern in both hemithoraces with visualization of the diaphragm or a corresponding curtain sign. An adequately diagnostic gastric ultrasound will be done in right lateral decubitus and demonstrate the liver in the near field, a great vessel (aorta or IVC) in the far field, and the stomach antrum deep to the liver in the near to mid-field with visualization of the hypo-echoic muscularis propria. These outcomes will be examined only in participants randomized to the Scan Group.
Rates of OR delays for optimization or further work-up. | From time of randomization to the time of interpretation of the last POCUS scan, assessed up to 2 weeks from randomization.
  Number of delays in the patient's surgery for optimization or further work-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hegazy, Assist. Prof, Principal Investigator — Schulich School of Medicine and Dentistry\Anaesthesia
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Canty DJ, Royse CF, Kilpatrick D, Williams DL, Royse AG. The impact of pre-operative focused transthoracic echocardiography in emergency non-cardiac surgery patients with known or risk of cardiac disease. Anaesthesia. 2012 Jul;67(7):714-20. doi: 10.1111/j.1365-2044.2012.07118.x. Epub 2012 Mar 27. PMID 22452367
- [Background] Heiberg J, El-Ansary D, Canty DJ, Royse AG, Royse CF. Focused echocardiography: a systematic review of diagnostic and clinical decision-making in anaesthesia and critical care. Anaesthesia. 2016 Sep;71(9):1091-100. doi: 10.1111/anae.13525. Epub 2016 Jun 27. PMID 27346556
- [Background] Canty DJ, Royse CF, Kilpatrick D, Bowyer A, Royse AG. The impact on cardiac diagnosis and mortality of focused transthoracic echocardiography in hip fracture surgery patients with increased risk of cardiac disease: a retrospective cohort study. Anaesthesia. 2012 Nov;67(11):1202-9. doi: 10.1111/j.1365-2044.2012.07300.x. Epub 2012 Sep 5. PMID 22950446